## PROTOCOL Protocol Submission Form

| Amendment | 1 |
|-----------------------------------------------------|----|
| Personnel Information | 1 |
| Subject Checklist | 4 |
| Study Location | 4 |
| General Checklist | 5 |
| Funding | 5 |
| Application Type Checklist | 6 |
| Exempt Paragraph(s) | 6 |
| Summary, Purpose, Procedures | 88 |
| Background and additional procedures | 10 |
| Subject Population (a-f) | 12 |
| Subject Population (g-k) | 13 |
| Recruitment Process, Subject Compensation and Costs | 13 |
| Risks | 15 |
| Benefits | 15 |
| Procedures to Maintain Confidentiality | 16 |
| Consent Information | 18 |
| Assent Background | 18 |
| HIPAA | 19 |
| Potential Conflict of Interest | 21 |
| Attachments | 22 |


Protocol # 21-05-6633 Date Printed: 08/22/2023

| Obligations | 23 |
|---------------|----|
| Event History | 24 |

C-PROTOCOL


Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

This Print View may not reflect all comments and contingencies for approval. **Important Note:** 

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

Decreased

#### \* \* \* Amendment \* \* \*

Amendment (1. Complete this one-page form, 2. Update the sections of your protocol that you are requesting to amend, 3. Electronically "sign" your application by clicking the check box on the Obligations page, 4. Remember to click "Submit Form" so that the IRB administrators receive your request.)

Summarize the proposed changes to the protocol in lay terms.

Updating language around data collection timeline, eligibility, and incentives to be more accurate.

Proceed to the appropriate section(s) of the protocol and make your changes.

IMPORTANT NOTE ON AMENDING ATTACHED DOCUMENTS: If you are requesting to amend a file that has been previously attached and approved, you MUST: 1. Delete the file that is currently attached, 2. Browse on your computer, and 3. Upload the revised file that you are requesting to use.

2. Indicate level of risk involved with the changes proposed.

(If level of risk has changed, please update the section 'Risks' in the protocol information.)

Increase X No Change Will you re-consent subjects.

3.

Approval Includes

List of sections (and questions) that have been changed/modified

\* \* \* Personnel Information \* \* \*

Starred items indicate required fields whenever that section is completed.

#### Principal Investigator

The University of Notre Dame defines "Investigator" as an individual who conducts a research study. If the study is conducted by a team of individuals, the Investigator is the responsible leader of the team. Name of Principal Investigator\* Degree (MD/PhD/BSN/etc.) PhD Cronin, Christopher Phone\* Email\* Fax 5746310427 ccronin1@nd.edu Research Department\* The University of Notre Dame Status | Mailing Address Check ALL that apply\* **Economics** Assistant Professor Faculty Staff

Postdoctoral Student

Graduate Student


Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

| | | Undergraduate<br>Student | | |
|---|---|---|---|---|
| | | Other | | |
| CITI training records are listed in the Training Details table below for accounts that have completed prerequisite courses and are affiliated with the University. If you do not have CITI training listed, please either manually enter your course information below, or go to the CITI Program website to confirm affiliation with the University. The Research Compliance Office will verify the last date of completion below. | | | | |
| CITI Training Date | | | | |
| <b>0</b> | | | ,,, | <u> </u> |
| Training Details | | | 1 | |
| Course | CourseCom | pletionDate | CourseID | EmailID |
| Human Research | 6/6/2016 2:3 | 32:28 PM 1 | | ccronin1@nd.edu |
| Human Research | 7/7/2021 3:4 | 19:41 PM 2 | ) | ccronin1@nd.edu |
| CITI Conflicts of Interest | 7/7/2021 4:1 | 3:46 PM 1 | | ccronin1@nd.edu |

#### **Faculty Advisor**

| Name of Faculty Advisor* | De | gree (MD/PhD/BS | SN/etc.) | Title |
|---|---|---|---|---|
| Email* | Ph | one | | Fax |
| Research Departmentfont * | | The University of Notre Dame Status Check ALL that apply* | | Mailing Address |
| | | Faculty | | |
| | | Staff | | |
| | | Postdoctoral Stu | dent | |
| | | Graduate<br>Student | | |
| | | Undergraduate S | Student | |
| | | Other | | |
| ALL research personnel are require years prior to engaging in any rese | ed to c | complete Human Selated activities. | Subject Research<br>So to CITI Progra | training from CITI within the last 2 m to complete. |
| The Research Compliance Office v | | | | |
| CITI Training Date | | - | Type of CITI training completed. | |
| | | | | · |

Other Investigator(s)

e-Protocol


Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

Degree (MD/PhD/BSN/etc.) Type of Investigator Name of Other Title Research Investigator Department Lieber, Ethan **Economics** Co-Investigator

#### **Study Coordinator**

| | Degree<br>(MD/PhD/BSN/etc.) | Title | Research Department |
|-----------------|-----------------------------|-------|---------------------|
| Tinoco, Brendan | | | |
| Perry, Brendan | | | |

#### **Administrative Contact**

| none | | |
|---|---|---|
| none | | |
| .0110 | | Fax |
| e University of Not<br>neck ALL that apply | re Dame Status | Mailing Address |
| Faculty | | |
| Staff | | |
| Postdoctoral Stud | dent | |
| Graduate<br>Student | | |
| Undergraduate St | tudent | |
| Other | | |
| complete Human S<br>related activities. G | ubject Research<br>o to CITI Prograi | training from CITI within the last 3 m to complete. |
| rify the last date of | completion below | v. |
| - | Type of CITI train | ning completed. |
| No training data i | is available | |
| 200 | Faculty Staff Postdoctoral Student Undergraduate S Other Omplete Human S elated activities. G fy the last date of | Staff Postdoctoral Student Graduate Student Undergraduate Student |

Other Personnel


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

| Name of Other Personnel | Degree<br>(MD/PhD/BSN/etc.) | Title | Research Department |
|---|---|---|---|
| Meghan Skira | | Associate Professor | |

\_\_\_\_\_\_

\* \* \* Subject Checklist \* \* \*

## **Subject Checklist**

#### Select All That Apply:

Economically/Educationally Disadvantaged

Elderly

X Healthy Adults

Homeless

Illiterate

Institutionalized Patients/Residents

Individuals with impaired decision-making capacity

Military Personnel

Minors (under 18)

Non-English Speakers

Persons incompetent to give consent (e.g., dementia, comatose, have legal guardians)

Pregnant women (Complete and attach the "Research Including Pregnant Women" Form that can be found in the resource library of our website: research.nd.edu)

Prisoners (Complete and attach the "Research for Including Prisoners" form that can be found in the resource library of our website: research.nd.edu)

Public Officials/Candidates for Public Office

Students (Elementary or secondary) (Upload a letter of agreement/permission from the schools.)

University Employees

University Students

X Other (please specify):

Mentally ill

\_\_\_\_\_\_

\* \* \* Study Location \* \* \*

#### **Study Location**

Select All That Apply - NOTE: Check "Other" and input text: 1.) If your study location is not listed, or 2.) If you would like to list details of your already-checked location (e.g., specific school within a school district)

University of Notre Dame Campus

X Local community

State-wide and/or Other States

Other University/College

Medical/Healthcare Facility

School(s)/School District(s)


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

------

Other (Specify)

Has this protocol been submitted to any other IRB?

N

Is this a multi-site project? (Different PIs at different institutions are conducting the same study or aspects of the same study.)

N

Will The University of Notre Dame function as the coordinating center or lead institution?

Υ

If Yes, upload a Multi-Site, Collaborative Research Form

If Yes and all institutions will review the research, upload IRB approval letters of letters of permission/support from the other sites (not under the jurisdiction of Notre Dame's IRB).

If yes and all institutions will be relying on a single IRB for review, upload a copy of the Reliance Agreement, signed by all institutions, to this application.

\_\_\_\_\_

\* \* \* General Checklist \* \* \*

#### **General Checklist**

#### Select All That Apply:

Administration of Dietary Supplements, substances or Other Chemicals (May be FDA-regulated)

Cancer patients or cancer tissues (Tissues requires Bio-Safety Committee approval)

Class Project

Human blood, cells, tissues, or body fluids (Requires Bio-Safety Committee approval)

Internet Research (Please complete and attach the Internet Research form that can be found in the resource library of our website: research.nd.edu)

Interview/Focus Group

Investigative Device (FDA-regulated)

IRB Authorization Agreement (IIA), Memorandum of Understanding (MOU), etc. (Upload a copy of the IIA or MOU)

Program Evaluation

X Protected Health Information (PHI) will be viewed, created, accessed, used, or disclosed.

HIPAA Authorization (Upload)

Waiver or Alteration of Authorization (Upload)

Activities Preparatory to Research (Upload)

X Limited Data Set and Data Use Agreement

Use and Disclosure of Decedents PHI without Authorization

Questionnaire/Survey

Request to Rely on another IRB (Upload a copy of the Reliance Agreement)

Research at Foreign Sites

Subject Pool (SONA).

Tissues to be sent out of this institution as part of a research agreement (Requires a Material Transfer Agreement (MTA))

Tissues to be stored for future research projects

Thesis or dissertation project

Use of Health Monitoring Equipment.

X Other

Impact Evaluation


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

\* \* \* Funding \* \* \*

NONE: This project does not have funding. (Please uncheck this selection to add a funding source)

Pending: This project is not currently funded, but a process for obtaining funds has been initiated. (Please add the anticipated funding source to the appropriate category below)

#### **Funding**

Add external and internal grant funding source(s) below: Federal Government, Other Gov. (i.e., State, local), Foundation or Other. Select "None" above if there is no external funding for the study.

#### **Notre Dame**

| Name of Funding Source | Proposal Number |
|-----------------------------------------------|-----------------|
| Wilson Sheehan Lab for Economic Opportunities | |

Funding for this study was secured by the Notre Dame Research Administration

\_\_\_\_\_

\* \* \* Application Type Checklist \* \* \*

#### Application type checklist

Not Human Subjects Research

X Exempt

Expedited/Full Board

-----

\* \* \* Exempt Paragraphs(s) \* \* \*

There are eight categories of research activities involving human subjects that may be exempt from the requirements of the Federal Policy for the Protection of Human Subjects (45 CFR 46). Select from the following applicable categories to determine if your research is exempt from expedited or full committee review. If your research qualifies under one or more of the exempt categories, proceed with the following application. If not, complete the expedited or full review application.

NOTE: The exempt categories below do not apply to research involving prisoners.

Select one or more of the following paragraphs applicable to your project:

- EDUCATIONAL PRACTICES: Research conducted in established or commonly accepted educational settings, involving normal
  educational practices that are not likely to adversely impact student's opportunity to learn required educational content of the
  assessment of educators who provide instruction. This includes most
  - i. Research on regular and special education instructional strategies; OR
  - ii. Research on the effectiveness of or the comparison among instructional techniques, curricula, or classroom management methods.

This category does not apply to use of school records of identifiable students or interviewing instructors about specific students.

2. EDUCATIONAL TESTS (COGNITIVE, DIAGNOSTIC, APTITUDE, ACHIEVEMENT), SURVEY PROCEDURES, INTERVIEW


Date Printed: 08/22/2023

Protocol # 21-05-6633

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

-----

## PROCEDURES,OR OBSERVATION OF PUBLIC BEHAVIOR(INCLUDING VISUAL OR AUDITORY RECORDING): Research involving these procedures is exempt, IF one of the following is correct:

- Any information obtained is recorded in such a manner that subjects CANNOT be identified, directly or through identifiers linked to the subjects; OR
- ii. Any disclosure of the subject's responses outside of the research could NOT reasonably place the subject at risk of criminal or civil liability or be damaging to the subject's financial standing, employability, educational advancement, or reputation; OR
- iii. Any information obtained is recorded by the investigator in such a manner that the identity of the human subjects CAN readily be identified, directly or through identifiers linked to the subjects, AND an IRB conducts a Limited IRB review to make the determination required by 45 CFR 46.111(a)(7)and the research is not subject to 45 CFR 46 Subpart D.

This exemption does not apply to children except for research involving observation of public behavior when the investigator does not interact with the children. Workplace meetings and activities, as well as classroom activities, are not considered "public behavior".

- X 3. RESEARCH INVOLVING BENIGN BEHAVIORAL INTERVENTIONS in conjunction with the collection of information from adult subjects through verbal or written response (including data entry) or audio visual recording, if the subject prospective agrees to the intervention and information collection, is exempt, IF
  - Any information obtained is recorded by the investigator in such a manner that the identity of the human subjects cannot readily be identified, directly or through identifiers linked to the subjects; OR
  - X ii. Any disclosure of the subject's responses outside of the research could NOT reasonably place the subject at risk of criminal or civil liability or be damaging to the subject's financial standing, employability, or reputation; OR
    - iii. Any information obtained is recorded by the investigator in such a manner that the identity of the human subjects can readily be identified, directly or through identifiers linked to the subjects, and an IRB conducts a Limited IRB review to make the determination required by 45 CFR 46.111(a)(7).
- X 4. EXISTING DATA: Secondary Research involving collection or study of existing data, documents, records, or biospecimens, for which consent is not required is exempt, IF:
  - i. The identifiable private information or identifiable biospecimens are publicly available; OR
  - ii. Information, which may include information about biospecimens, is recorded by the researcher in such a manner that subjects cannot be identified, directly or through identifiers linked to the subjects, the investigator does not contact the subjects, and the investigator will not re-identify the subjects; OR
  - X iii. The research involves only information collection and analysis involving the investigator's use of identifiable health information when that use is regulated under 45 CFR parts 160 and 164, subpart A and E, for the purposes of "health care operations" or "research" as those terms are defined at 45 CFR 164.501 or for "public health activities and purposes" as described under 45 CFR 1.512(b); OR
    - iv. The research is conducted by, or on behalf of, a Federal department or agency using government-generated or government-collected information obtained for non-research activities, if the research generates identifiable private information that is or will be maintained on information technology that is subject to and in compliance with section 298(b) of the E-Government Act of 2002, 44 U.S.C. 3501 note, if all of the identifiable private information collected, used, or generated as part of the activity will be maintained in systems of records subject to the Privacy Act of 1974, 5 U.S.C. 5521, and, if applicable, the information used in the research was collected subject to the Paperwork Reduction Act of 1995, 44 U.S.C. 3501et seq.
  - RESEARCH AND DEMONSTRATION PROJECTS CONDUCTED BY OR SUBJECT TO THE APPROVAL OF DEPARTMENT OR AGENCY HEADS: This research is exempt IF it is designed to study, evaluate, or otherwise examine:
    - Public benefit or service programs;
    - ii. Procedures for obtaining benefits or services under those programs;OR
    - iii. Possible changes in or alternatives to those programs, OR
    - Changes in methods or levels of payment for benefits or services under those programs.

Such projects include, but are not limited to, internal studies by Federal employees, and studies under contracts of consulting arrangements, cooperative agreements, or grants. Exempt projects also include waivers of otherwise mandatory requirements using authorities such as sections 1115 and 115A of the Social Security Act, as amended.

Note: Each Federal department or agency conducting or supporting research [post on Website]


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

-----

- TASTE AND FOOD QUALITY EVALUATION AND CONSUMER ACCEPTANCE STUDIES: This research is exempt, IF:
  - i. Wholesome foods without additives are consumed; OR
  - ii. A food is consumed that contains a food ingredient at or below the level and for a use found to be safe by the Food and Drug Administration (FDA) or approved by the Environmental Protection Agency (EPA) or the Food Safety and Inspection Service (FSIS) of the US Department of Agriculture (USDA); OR
  - iii. A food is consumed that contains an agricultural chemical or environmental contaminant at or below the level found to be safe by the FDA or approved by the EPA or the FSIS of the USDA.
- 7. STORAGE OR MAINTENANCE OF INFORMATION FOR SECONDARY RESEARCH FOR WHICH BROAD CONSENT IS REQUIRED: The protocol is eligible for exemption if:
  - It involves storage or maintenance of identifiable private information or identifiable biospecimens for secondary research use; AND
  - ii. All the identifiable information or identifiable biospecimens that are to be stored and/or maintained for secondary research have been or will be collected for another "primary" purpose; AND
  - iii. Broad consent for the storage or maintenance of their identifiable information or identifiable biospecimens for secondary research use will be obtained from ALL subjects; AND
  - iv. The protocol does not include any activities that do not qualify for exemption; AND
  - v. The protocol is not for an FDA regulated clinical investigation; AND
  - ri. The IRB conducts a Limited IRB Review and makes the determinations required by 45 CFR 46.111(a)(8)
- SECONDARY RESEARCH FOR WHICH BROAD CONSENT IS REQUIRED: Research involving the use of identifiable private
  information or identifiable biospecimens for secondary research use is eligible for exemption, if the following criteria are met:
  - Broad consent for the storage, maintenance, and secondary research use of the identifiable private information or identifiable biospecimens was obtained in accordance with 45 CFR 46.116(a)(1) through (4), (a)(6), and (d); AND
  - ii. Documentation of informed consent or waiver of documentation of consent was obtained in accordance with 45 CFR 46.117; AND
  - iii. An IRB conducts a Limited IRB review and makes the determination required by 45 CFR 46.111(a)(7) and makes the determination that the research to be conducted is within the scope of the broad consent referenced in paragraph (d)(8)(i) of this section; AND
  - iv. The investigator does not include returning individual research results to subjects as part of the study plan. This provision does not prevent an investigator from abiding by any legal requirements to return individual research results.

\_\_\_\_\_

\* \* \* Summary, Purpose, Procedures \* \* \*

Title (Please indicate if the protocol title is different from the proposal title)

Recovery Resource Council - Veteran Incentives

# This submission is a renewal of already-approved research using the new protocol submission form

Proposed Start Date:\* 09/01/2021 Proposed End Date:\* 09/02/2024

- Summary
- a) Provide a brief summary of the scope of work of this project, using non-technical terms that would be understood by a non-scientific reader. This summary should be no more than 200 words.

Recovery Resource Council (RRC) is one of the largest and most comprehensive non-profit mental and behavioral healthcare providers in North Texas. Accredited by the Joint Commission in Behavioral Health and licensed by the State of Texas as an Outpatient Treatment Center, RRC strives to promote wellness and recovery from alcohol and substance use disorders and trauma. An important component of RRC programming is providing free counseling services to hundreds of U.S. veterans who struggle with mental health issues such as PTSD and severe depression annually. While RRC observes great success for veterans who complete


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

\_\_\_\_\_\_

mental health issues such as PTSD and severe depression annually. While RRC observes great success for veterans who complete counseling, attendance can be a major obstacle.

RRC and the Wilson-Sheehan Lab for Economic Opportunities (LEO) are partnering to explore an experimental research study that will generate evidence on the impact of incentivizing veterans to complete a series of prescribed counseling sessions on session attendance and completion rate. To do this, RRC will offer financial incentives of \$500 to every client who completes a group of 6 counselling sessions, for up to 18 sessions and \$1500. The research team will evaluate the impact and cost-effectiveness of the therapy incentives via a randomized controlled trial.

LEO will conduct this evaluation using administrative data from RRC, the Ray Marshall Center at the University of Texas at Austin, and the VA.

#### 2. Purpose

a) Describe the purpose for the proposed project as well as the hypotheses/research questions to be examined.

This research project will investigate the impact of RRC's therapy incentives on veterans' counselling session attendance and completion rates by evaluating differences in outcomes between the group offered incentives and the control group. The research question to be tested is, "What is the effect of incentivizing veterans to persist with prescribed counselling sessions on completion rate and on total sessions attended?"

b) What do the investigators hope to learn from this project?

Investigators hope to learn whether financial incentives like those offered by RRC are an effective way to improve veterans' counselling session attendance and completion rates. Due to the program specific focus of this research, results from this evaluation will also be valuable for RRC operations. If, for instance, evidence shows incentivization to be effective for improving these outcomes, RRC will be better positioned to expand the program and serve more individuals. In addition to RRC, the results from this research could have implications for similarly targeted programs elsewhere.

#### Procedures

a) Describe in chronological order of event(s) how the activities will be conducted, providing information about all procedures (e.g. interventions/interactions with subjects, data collection, photographing, audio and video recording), including follow up procedures.

We propose to evaluate the impact of RRC's therapy incentives using a randomized control trial research design.

- 1.Veterans who are referred to RRC are subject to an eligibility screening via phone, during which time they must ensure that they are a veteran. Eligible veterans are then assigned an intake session time, during which they show any requested documentation, complete an intake form, complete an initial mental health assessment, and go through the informed consent process with RRC staff. Any participant who does not want to participate in the study will still receive all services as usual. After a participant gives consent, they are enrolled in the study. Randomization will be done virtually, so that results can be communicated to veterans immediately during their intake session.
- 2. The treatment group will be informed that if they attend their first six counselling sessions, they will be given a \$500 gift card. If it is determined that they need more sessions, they will be given the same incentive to attend 6 more sessions. The same process continues again after the completion of 12 sessions. The content of all counseling sessions will not be impacted by the designation of treatment or control group.
- 3. Those in the control group will receive "business as usual" services offered by the RRC, which includes the same counseling services and evaluation of how many sessions an individual is recommended to receive.
- 4. Administrative data will be periodically collected from the various data partners in line with the pending data sharing agreements.
- 5. LEO and the Ray Marshall Center at the University of Texas at Austin and the VA will sign Data Sharing Agreements to facilitate the study of therapy incentives on veteran outcomes.
- Be sure to identify what procedures are experimental and what are standard of care or established practice for the condition/situation.

The experimental portion of these procedures is the random assignment of individuals to be offered or to not be offered financial incentives for therapy. The established practices for this process include the data sharing procedures described previously, which are conducted to protect client information. Other than informing individuals of the gift cards, then reassessing and re-informing them of potential additional financial incentives, and including an informed consent process and collecting some additional personal information in an online form, counselling services itself will not change as a result of this study. Individuals who are not offered the opportunity for therapy incentives will have access to the normal counseling services provided by RRC staff.


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

------

Importantly, the control group (individuals who are randomly selected to not receive re-entry programming) will not be created solely for the study. There are more therapy incentive-eligible individuals within the community than RRC has the resources to serve. Consequently, RRC has agreed to offer therapy incentives through a lottery-based system, under which eligible individuals will be randomly assigned to either the treatment group or the control group.

b) Explain who will conduct the procedures and where and when they will take place. Indicate the frequency and duration of visits/sessions as well as the subject's total time commitment for the study. Include how the data will be collected (i.e. in person or online).

The RRC staff member who is working with the client during intake will be in charge of going through the informed consent process during the preliminary intake session using the online Qualtrics survey form. The staff member will read through the consent information and then ask potential participants a mandatory question of if they consent to research or not. After a participant gives consent, they are enrolled in the study. Randomization will be done virtually via the survey form, so that results can be communicated to veterans during their intake session.

Services will take place at the RRC locations in Fort Worth, Dallas, and Denton, Texas. For those who are randomly selected to the control group, there is no additional time commitment imposed by the study beyond the informed consent process.

 Indicate that the instruments used are in the public domain or provide appropriate documentation of permission to use each scale.

Not applicable.

c) For school-based activities where class time is used, describe in detail the activities planned for non-subjects and explain where both subjects and nonsubjects will be located during the activities.

Not applicable.

d) State if deception will be used. If so, provide a rationale and describe debriefing procedures. Submit a debriefing script in attachments section

Deception will not be used.

- e) Do any of the following apply.
  - i. Will subjects be audio recorded?

N

ii. Will subjects be videotaped?

IN

iii. Will subjects be photographed?

Ν

If yes to i, ii or iii, explain the collection process and use in the context of this research of such media

f) Will the proposed research involve the use of existing data/specimens? If yes, please check all that apply:

Ν

- i. The research involves data from publicly available sources
- ii. That data will be recorded by the investigator in such a manner that subjects cannot be identified.
- iii. Any link to identifying information has been destroyed

#### \* \* \* Background and additional procedures \* \* \*

- 4. Background and additional procedures
- a. Relevant Background: Discuss the present knowledge, appropriate literature and rationale for conducting the research. Include the rationale for the selected subject population.

Studies indicate that many individuals suffering with mental health difficulties often fail to obtain and complete adequate mental health treatment (Swift & Greenberg, 2012; Wierzbicki & Pekarik, 1993). Low therapy initiation, low attendance, and premature discontinuation are persistent areas of concern in spite of the effectiveness of trauma-focused therapy treatments. Premature discontinuation of psychotherapy, in particular, poses a significant barrier to treatment efficacy for both clients and healthcare providers. Individuals who prematurely drop out of therapy have generally been found to experience poorer treatment outcomes (Cahill et al., 2003; Lampropoulos, 2010; Pekarik, 1992). With respect to veterans specifically, recent studies of PTSD treatment

e-Protocol


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

\_\_\_\_\_\_

(Cahill et al., 2003; Lampropoulos, 2010; Pekarik, 1992). With respect to veterans specifically, recent studies of PTSD treatment programs have found that many veterans who enter treatment do not stay for the intended treatment length and do not achieve clinical benefits (Hoge et al., 2014; Mott et al., 2014; Watts et al. 2014). At the same time, fewer missed sessions and overall treatment completion have been associated with better treatment outcomes for veterans (Rutt et al., 2018; Tarrier et al., 2000). Research studying self-reported reasons for premature discontinuation among veterans cites reasons including issues with scheduling, logistical barriers, and length of therapy, and concerns with therapy efficacy (Brown et al., 2017).

There is growing interest in using financial incentive schemes to promote positive habit formation in both health and non-health related contexts. Research studies have focused on incentivized behaviors in a range of health-related programs, including smoking cessation (Volpp et al. 2009), exercise (Charness & Gneezy, 2008), and workplace wellness (Jones et al., 2019; Rief et al., 2020). Some such studies have found positive relationships between incentives and desired health changes; for example, an analysis of studies on voucher-based reinforcement therapy (VBRT) for substance use disorders found that in general, VBRT generated better outcomes in comparison to control groups (Lussier et al., 2005). In particular, a study implementing a progressively lowered pay scale rewarding therapy attendance and retention shows that these discounted fee incentives are associated with improved clinical functioning (Stanley et al., 2016).

We conclude that it is relevant to understand how we can address the issues of retention and completion in veteran therapy and ensure that veterans suffering with mental health difficulties complete adequate mental health treatment. Evaluating the RRC therapy incentive intervention, which offers potential encouragement for veterans to attend and complete counselling sessions, would improve our current knowledge about the effectiveness of such programming.

b. Describe the statistical methods of the research and plans for analysis of the data (i.e. planned statistics, justification of sample size, etc.).

Following the construction of this study as a randomized control trial, those assigned to treatment and control groups should look equivalent to each other on average. Thus, any difference in outcomes between the two groups could be attributed to their treatment status. After individuals have been randomized into these groups and the study begins, LEO will monitor outcomes into the future and compare them.

In particular, relevant outcomes will be compared with a statistical model that estimates the average difference in outcomes between those that are assigned to the treatment and control groups.

To reduce residual variance we plan to estimate the differences in outcomes using an Ordinary Least Squares (OLS) model. Specifically, we will estimate the following intent-to-treat (ITT) model:

yi =β0 + Tiβ1 + xiβ2 + εi

where yi is an indicator for key outcome variables, such as the number of counselling session attended, and xi represents a vector of observed characteristics for person i. The variables in x will include demographic characteristics such as age, age squared, categorical race indicators, indicators for ethnicity and gender. The key covariate in the analysis will be the dummy variable, Ti, which equal 1 if the respondent is assigned to the treatment group (i.e. offered to participate in the re-entry program) and zero otherwise.  $\epsilon$ i is an error term. We will measure the outcomes every year after randomization, determining short-term, mid-term, and long-term effects of the program. Treatment-on-the-treated (TOT) effects will be estimated via an instrumental variable (IV) model, using assignment to treatment as an instrument for participation in the program. Program participation (or take-up) is defined as attending the first day of programming.

- c. Alternative Procedures. Describe any alternatives to participating in the research. (e.g., standard of care treatment, etc.). Any standard treatment that is being withheld must be disclosed. This information must be included in the consent form.
- d. Will subjects be followed after their active participation is complete?

If yes, explain why and describe how:

e. Will subjects have access to the study treatment/procedure after completing the study? If yes, explain why and describe how:

(Explicit consent must be obtained for use of these methods for Expedited and Full Board studies.)


Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives **Protocol Type:** Protocol Submission Form **Date Submitted:** 08/14/2023 This Print View may not reflect all comments and contingencies for approval. **Important Note:** Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. \* \* \* Subject Population (a-f) \* \* \* Subject Population 5. a) How many subjects to you intend to enroll and/or how many subject records to you intend to access? At this site # of subjects # of records ii. At all sites N/A # of subjects # of records Inclusion and Exclusion Criteria (e.g., Participants must have 20/20 vision, Participants must be 30-45 years of age, etc.) b) Identify inclusion criteria. Eligibility Criteria: Voluntarily agree to participation requirements outlined in the informed consent form
 18 years of age or older Holds veteran status Possesses and is willing to share SSN
 Possesses and is willing to share an active email address
 Is participating in individual (not family) counseling Outside of existing referrals, little to no formal study recruitment will be needed because veterans will be informed of and enrolled in the study during their intake session that begins their relationship with RRC. Currently, veterans are referred to RRC by the VA, as well as by friendly agencies, word of mouth, and community partners. ii. Identify exclusion criteria. Individuals who do not meet the eligibility requirements above will be excluded. Individuals who are not interested in participating will be excluded, as well as individuals who do not consent. What is the rationale for studying the requested group(s) of participants? c) Primarily, the criteria described above are set by RRC. The veteran therapy incentives program is an intervention designed to improve counselling session attendance and completion rates for veterans. Thus, the rationale for studying this group of participants is that we would like to examine whether the therapy incentives program is an effective means to improve outcomes of veterans in the North Texas community. d) If women, minorities, or minors are intentionally excluded, a clear compelling rationale must be provided. Examples for N/A not including minors: disease does not occur in children; drug or device would interfere with normal growth and development; etc. State if any of the subjects are students, employees, or laboratory personnel. Please explain how subjects will be N/A e) protected from coercion and undue influence Please describe the expertise you have, or have access to, which prepares you to conduct research in this location and/or with this subject population, including specific qualifications (e.g., relevant coursework, background, experience, and training). Also, explain your knowledge of local community attitudes and cultural norms and cultural sensitivities necessary to carry out the research (e.g., differences with U.S. culture). f)


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

-----

| * * * Subject Population | (q-k) | * | * | * |
|--------------------------|-------|---|---|---|
|--------------------------|-------|---|---|---|

- 5. Subject Population (Input N/A if not applicable)
- g) Will bilingual or multilingual subjects be recruited?
- h) Will non-English speaking subjects be recruited?

Ν

If yes, state language(s) spoken (other than English):

i) Will subjects be less than 18 years of age?

Ν

- Describe any planned screening procedures. Attach your screening document(s) (e.g., health history questionnaire) in the Attachment Section (#16).
- k) Will you be conducting international/transnational research and enrolling participants at foreign sites?

Ν

\_\_\_\_\_

## \* \* \* Recruitment Process, Subject Compensation and Costs \* \* \*

- 6. Recruitment Process:
- a) Describe the step-by-step procedures for identifying and recruiting potential research subjects or requesting pre-existing data or materials.
  - List any specific agencies or institutions that will provide access to prospective subjects.
  - Identify who will contact prospective subjects and how.
  - 1.Veterans who are referred to RRC for mental health services will complete an eligibility screen over the phone, during which time they will confirm their veteran status.
  - 2. Eligible veterans are then assigned an intake session time, during which they show any requested documentation, complete an intake form, complete a baseline mental health assessment, and go through the informed consent process with RRC staff. All clients are given a case ID during the intake session. During this session, the RRC staff member working with the client during intake will be responsible for enrolling the individual into the study, should they provide consent. Enrollment and consent procedures will be conducted using the online Qualtrics survey form. Any participant who does not want to participate in the study will still receive all services as usual.
  - 3.After collecting consent from participants, individuals will be randomly assigned to either the treatment or control group during their intake meeting. Randomization will be done virtually via the survey form, so that results can be communicated to veterans immediately during their intake session.
  - 4.The start of the intervention entails RRC intake staff informing veterans in the treatment group that they will receive a \$500 gift card upon completing the first 6 sessions. It is not until the first 6 sessions are completed that gift card will be distributed to treated individuals and they will be re-assessed to determine if they need another 6 sessions. Other than informing individuals of the money and then re-assessing and re-informing them of potential additional financial incentives, participants will receive the normal counseling services provided by RRC staff.
  - 5. Those in the control group will receive "business as usual" services offered by the RRC, which includes the same counseling services and evaluation of how many sessions an individual is recommended to receive.
- b) Planned Subject Identification Methods:

N/A

Direct advertising

c)

7.

a)

b)

c)

d)

e)

not wish to participate in the study.

Not applicable.

# PROTOCOL Protocol Submission Form

Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Submission Form Protocol Title:** Recovery Resource Council - Veteran Incentives **Protocol Type:** Protocol Submission Form **Date Submitted:** 08/14/2023 This Print View may not reflect all comments and contingencies for approval. **Important Note:** Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Chart/database review Living conditions (e.g., nursing home residents) From PI's own practice/clinic Class participants Circumstance (e.g., homelessness) X Referrals The University of Notre Dame Subject Pool Organization mailing lists Other (please specify): Planned Recruitment Materials/Methods: X N/A Flyers/posters Phone Scripts Letters to providers/schools/organizations Television ads Newspaper ads Letters to prospective subjects Radio ads **Oral Scripts** PowerPoint presentations Internet ads/postings Fmail Face to face interactions The University of Notre Dame Subject Pool Other (please specify): (All advertising must be submitted for review in its final printed/recorded form) Note: Attach copies of ALL recruitment materials in the attachment Section **Subject Compensation and Costs:** Will subjects receive compensation for participation? Total amount (in dollars or equivalent) 500 Form of Compensation: Raffles/lotteries Cash Check Course/extra credit X Gift card/certificate Reimbursement only Voucher Other (please specify) Describe the remuneration plan (Include when subjects will be paid, whether payment will be prorated and whether a 1099 will be issued.) Subjects have a 50/50 chance of being placed in the treatment group (the randomization procedure described elsewhere determines treatment status). Every subject in the treatment group will be informed that those who complete 6 counselling sessions will be issued a \$500 gift card payment, received immediately after the 6th session is completed. During the 5th session, the individual will be reassessed to determine if they need an additional 6 sessions. If so, they will be informed of further financial incentives at this time (i.e., at the end of the 5th session). If the subject attends the additional 6 sessions, then they will be issued another \$500 gift card payment (i.e., at the conclusion of the 12th session) and the process will be repeated one final time. After these 18 sessions there will be no further financial incentive, thus the maximum amount that can be awarded to one individual is \$1500. Gift card payments are distributed by the partner organization and thus any tax obligations are the partner organization's responsibility. They are currently in contact with their auditor to determine what forms need to be filed. For raffles include the number of prizes, nature and value of each prize. Not applicable. If extra course credit is offered be sure to address the alternative means by which students can accrue extra course credit should they


Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives **Protocol Type:** Protocol Submission Form **Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

| | If yes, explain: |
|---|---|
| \M/bo io | responsible for costs incurred due to injury/harm? |
| VVIIO IS | responsible for costs incurred due to injury/namir |
| | * * * Risks * * * |
| Risks | (Input N/A if not applicable) |
| exposed<br>iny rese | artment of Health & Human Services (HHS) Regulations define a subject at risk as follows: "any individual who may be I to the possibility of injury, including physical, psychological, or social injury, as a consequence of participation as a subject earch, development, or related activity which departs from the application of those accepted methods necessary to meet his or which increases the ordinary risks of daily life, including the recognized risks inherent in a chosen occupation or field of |
| PI's ev | aluation of the overall level of Risk. (Please check one: minimal or minimal.) |
| Mini | imal (everyday living) |
| | imal (everyday living)<br>nimal (greater than everyday living) |
| Min<br>Descril<br>invasion | · |
| Describinvasion each reach between | himal (greater than everyday living) be all known risks or discomforts associated with study procedures whether physical, psychological or social (e.g., pain, strong of privacy, breach of confidentiality) noting probability and magnitude of potential harm. Specify the risks(s) associated vesearch procedure or test. ey risk is the possible invasion of privacy of a subject or family, including the use of personal information or records. The risk of confidentiality of any private or personal information collected during the course of the study is unlikely. All files transfer |
| Descril invasion each reach between identifications. | be all known risks or discomforts associated with study procedures whether physical, psychological or social (e.g., pain, strong of privacy, breach of confidentiality) noting probability and magnitude of potential harm. Specify the risks(s) associated versearch procedure or test. Bey risk is the possible invasion of privacy of a subject or family, including the use of personal information or records. The risk of confidentiality of any private or personal information collected during the course of the study is unlikely. All files transferent he study partners will be transferred by secure web transfer services, encrypted and password protected in transit. Any fiable information will be coded and stored separately from de-identified analysis files. Be the procedures or safeguards in place to protect against or minimize potential risks (e.g., referral to psychological counse) |
| Mirr Descrii invasic each reference to the key between identified to the control of the control | be all known risks or discomforts associated with study procedures whether physical, psychological or social (e.g., pain, strong of privacy, breach of confidentiality) noting probability and magnitude of potential harm. Specify the risks(s) associated versearch procedure or test. Bey risk is the possible invasion of privacy of a subject or family, including the use of personal information or records. The risk of confidentiality of any private or personal information collected during the course of the study is unlikely. All files transferent he study partners will be transferred by secure web transfer services, encrypted and password protected in transit. Any fiable information will be coded and stored separately from de-identified analysis files. Be the procedures or safeguards in place to protect against or minimize potential risks (e.g., referral to psychological counse) |
| Descrilinvasion each receptive identification. Descriling Descriling Descriling Properties out of the control | be all known risks or discomforts associated with study procedures whether physical, psychological or social (e.g., pain, stand privacy, breach of confidentiality) noting probability and magnitude of potential harm. Specify the risks(s) associated varies arch procedure or test. By risk is the possible invasion of privacy of a subject or family, including the use of personal information or records. The rist of confidentiality of any private or personal information collected during the course of the study is unlikely. All files transferent he study partners will be transferred by secure web transfer services, encrypted and password protected in transit. Any fiable information will be coded and stored separately from de-identified analysis files. By the procedures or safeguards in place to protect against or minimize potential risks (e.g., referral to psychological course cos). By the procedures or safeguards in place to protect against or minimize potential risks (e.g., referral to psychological course cos). By the procedures or safeguards in place to protect against or minimize potential risks (e.g., referral to psychological course cos). By the procedures or safeguards in place to protect against or minimize potential risks (e.g., referral to psychological course cos). By the procedures or safeguards in place to protect against or minimize potential risks (e.g., referral to psychological course cos). By the procedures or safeguards in place to protect against or minimize potential risks (e.g., referral to psychological course cos). By the procedures or safeguards in place to protect against or minimize potential risks (e.g., referral to psychological course cos). By the procedure or definition or records. The risks (e.g., referral to psychological course cos). By the procedure or definition or records. By the risks (s) associated visit risks (e.g., referral to psychological course cos). By the procedure or definition or records. By the risks (s) associated visit risks (e.g., referral to psychologic |
| Descril invasic each re The ke breach to betwee identifing the period of | be all known risks or discomforts associated with study procedures whether physical, psychological or social (e.g., pain, ston of privacy, breach of confidentiality) noting probability and magnitude of potential harm. Specify the risks(s) associated besearch procedure or test. by risk is the possible invasion of privacy of a subject or family, including the use of personal information or records. The rish of confidentiality of any private or personal information collected during the course of the study is unlikely. All files transferent he study partners will be transferred by secure web transfer services, encrypted and password protected in transit. Any inable information will be coded and stored separately from de-identified analysis files. be the procedures or safeguards in place to protect against or minimize potential risks (e.g., referral to psychological counsels). orting statistical results, only aggregate statistics like regression coefficients and sample/subsample means will be reported fore, readers will not be able to identify individual respondents from published work. ata stored at the University of Notre Dame will be stored on our secure CorpFS servers. Only members of the research teams access to the folders containing secure data through an access control list. Data is only accessible when logged into the staff Confidentiality Agreement, agreeing to access data only for the purpose of the research project. Data cannot sed unless authorized users are logged in with their authenticated username/password combination through the two-step is the staff confidentiality agreement, agreeing to access data only for the purpose of the research project. Data cannot sed unless authorized users are logged in with their authenticated username/password combination through the two-step is the research project. |

\* \* \* Benefits \* \* \*


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Direct benefits to subjects (if applicable)

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

\_\_\_\_\_

#### 9. Benefits

a) Discuss any potential benefits that would justify involvement of subjects in this study.

ii. Indirect benefits to society

b) Explain how the potential benefits justify the potential risks involved in participation in this research.

\_\_\_\_\_\_

\* \* \* Procedures to Maintain Confidentiality \* \* \*

## 10. Procedures to Maintain Confidentiality

Which of the following types of data will you work with:

#### X Identifiable

Information is considered to be identifiable when it can be linked to specific individuals by the investigator(s) either directly or indirectly through coding systems, or when characteristics of the information obtained are such that by their nature a reasonably knowledgeable person or investigator could ascertain the identities of individuals. Therefore, even though a dataset may have been stripped of direct identifiers (names, addresses, student ID numbers, etc.), it may still be possible to identify an individual through a combination of other characteristics (e.g., age, gender, ethnicity, and place of employment).

Explain why you could not complete the research using de-identified data.

Use of identifiable data (first and last name, SSN) is essential to link RRC records to data provided by the Ray Marshall Center (RMC) and the VA, which will be used to track mid- to long-term outcomes of the study such as employment and earnings.

#### Anonymous

Data are anonymous if no one, not even the researcher, can connect the data to the person who provided it—no identifying information is collected from the individual. Investigators must be aware, however, that even if no direct identifiers (name, address, student ID, etc.) are collected, identification of a participant may be possible from unique individual characteristics (indirect identifiers). For example, a participant who is a member of a certain ethnic group or who was studied because of distinctive personal accomplishments or medical history might be identifiable from even a large data pool.

#### De-identified

If the dataset has been stripped of all identifying information and there is no way that it could be linked back to the subjects from whom it was originally collected (through a key to a coding system or by any other means). Note: This also applies if the source of the data is identifiable but the data collected is not.

#### Coded

This refers to data that have been stripped of all direct subject identifiers, but in this case each record has its own study ID or code, which is linked to identifiable information such as name or medical record number. The linking file must be separate from the coded data set. This linking file may be held by someone on the study team (e.g. the PI) or it could be held by someone outside of the study team (e.g. researcher at another institution). A coded data set may include limited identifiers under HIPAA. Of note, the code itself may not contain identifiers such as subject initials or medical record number.

a) If information derived from the study will be provided to the subject's personal physician, a government agency, or any other person or group (other than the research team), describe to whom the information will be given and the nature of the information, if applicable.

The Ray Marshall Center (RMC) at the VA are agencies with which we are interested in linking client information with in order to learn about outcomes of interest, including future earnings (RMC) and hospitalizations (VA). Via coordination with RRC, these agencies will be provided with the minimum amount of client information required for them to identify individuals within their own records. After being linked to outcomes of interest, data will be stripped of personally identifiable information.

C-PROTOCOL


Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

This Print View may not reflect all comments and contingencies for approval. **Important Note:** 

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

b)

Explain how you will protect subjects' privacy.

Note: Privacy refers to persons and their interest in controlling the access of others to themselves. For example, based on their privacy interest's people want to control:

- The time and place where they give information.
- The nature of the information they give.
- The nature of the experiences that are given to them.
- Who receives and can use the information.

For example, persons might not want to be seen entering a place that might stigmatize them, such as a pregnancy-counseling center that is clearly identified as such by signs on the front of the building. Please keep this definition in mind as you respond to this item.

Program services will take place at the RRC locations in Forth Worth, Dallas, and Denton, Texas as usual. The study will not introduce any additional public exposure.

c)

Describe how you will maintain the confidentiality of subjects' information.

Note: Confidentiality pertains to the treatment of information that an individual has disclosed in a relationship of trust and with the expectation that it will not be divulged to others (without permission) in ways that are inconsistent with the understanding of the original disclosure. Please keep this definition in mind as you respond to this item.

Only approved individuals who have undergone human subjects certification and who are listed on the approved IRB protocol have access to relevant datasets.

Data are transported between RRC and the Notre Dame HIPAA compliant system using a secure File Transfer Portal (sFTP) or equivalent. The secure portal automatically includes the following security measures at a minimum: Encryption – All files are transferred with 256 bit FIPS encryption.

Authentication - All downloads are authenticated, ensuring that only the intended recipient will receive the files.

Log – All transfers are logged, giving proof of any files sent in or out of the secure system. Scanning – All files are Virus Scanned when transferred and deleted if found to be infected.

Blocked Extensions – File types most commonly used to spread viruses are blocked.

LEO handles PHI according to all standards and procedures outlined by the Health Insurance Portability and Accountability Act of 1996 (HIPAA), and the subsequent Privacy Rule of 2002 and Security Rule of 2003. All sensitive digital data at CEHI reside within a limited access, secure, HIPAA compliant network on cloud based servers where all access to data requires using dual authenticated credentials to ensure that data are inaccessible to unauthorized users. The system is housed in the University of Notre Dame's Amazon Web Services (AWS) infrastructure.

LEO will store the data in the cyberinfrastructure that is part of the Compliant Cloud Computing for PHI (C3PHI) environment. C3PHI exists within an AWS Virtual Private Cloud (VPC) which provides a secure isolated network environment. C3PHI is connected to a network isolated ND Shared Services VPC which provides security services such as system monitoring, identity management, remote resource provisioning, critical security patch repositories and system/data transit logging. Identity management is provided to remote users via Okta and internally within the VPCs via Active Directory. Both the C3PHI and ND PHI Shared Services VPC are instantiated with AWS Cloud Formation scripts based on AWS templates to meet HIPAA best practices. The VPCs are isolated from the number and accessible only via the authorization tools meetinged. the public internet and accessible only via the authentication tools mentioned.

Within C3PHI, Windows workstations and support servers are provisioned (and patched) using both AWS EC2 instances and AppStream technology. All of the Windows systems are secured using the Microsoft Security Compliance Manager (SCM). This method provides Desired Configuration Management (DCM) templates based on Microsoft Security Guide recommendations and industry best practices to ensure high security, prevent configuration drift, and ensure compliance. AppStream environments are transient, retaining only user-specific configuration changes, such as apps pinned to the start bar, from session to session. They are reset to stock configuration at the start of each new session, and any locally-stored data is erased.

Data is provisioned to the workstation via secure SMB interfaces to AWS S3 storage buckets. AWS S3 storage allows for higher resolution logging of individual file movements and accesses. Users access the system via a browser session where no data can be transferred between the user's local desktop and the remote workstation. Data transfers out of the system must be done through a data transfer node managed by authorized system administrators and lab managers. Users can place data within C3PHI into a transfer node; but only the authorized data managers can retrieve data from the secure transfer node onto local systems outside of the secure C3PHI environment.

Users access the data via secure (patched), firewalled computers and encrypted VDI sessions. All original files, as well as all working and temporary files remain only on computers that are part of this secure network. This system may be upgraded as time and technology advance.

All storage and analysis of data take place exclusively in the secure C3PHI environment.

e-Protocol


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

-----

d) Who will have access to study records or specimens? (Please identify specific team members by name.)

Pls: Christopher Cronin, Ethan Lieber, and Meghan Skira. LEO Staff: Maura Hogaboom.

e) If you plan to use existing data, records or specimens, what is the source of the data/records/specimens, and how will you access them?

NOTE: "Existing" means data or specimens collected (i.e., on the shelf) prior to the IRB application submission. It includes data or specimens collected for research and non-research activities.

Not applicable.

f) How will subjects be asked to provide their permission for release of identifiable data collected as a part of this proposed research (e.g., pictures, recordings, responses to research questions), now or in future? Explain and include appropriate statements in consent materials.

Participants will be informed of the research study during the informed consent process.

g) If using existing data/biological specimens, will the researchers have access to a code linking the data to personally identifiable information?

Not applicable.

h) If the data is coded, explain where the key to identifiers will be stored, how it will be protected, and who will have access to it.

Not applicable.

i) Explain why, where, in what format, and for how long data/specimens will be retained.

Data will be maintained for the length of the study. Data will be stored in .csv and .dta files in a secure HIPAA-compliant environment at the University of Notre Dame.

\_\_\_\_\_

\* \* \* Consent Information \* \* \*

#### 11. Consent Information

11 a & b only apply to exempt applications

a) How will subjects be informed of procedures, intent of the study, and potential risks to them?

Subjects will be informed of procedures, intent, and risks during the informed consent process.

b) How will subjects be informed they may withdraw at any time without penalty?

Subjects will be informed that they may withdraw at any time without penalty during the informed consent process.

Note: Attach, in the Attachments Section, written and/or verbal instructions the subject will receive.

Please provide consent process background information below.

#### Informed Consent

| Title | Consent Type | Attached Date | Submitted Date |
|------------------|------------------|---------------|----------------|
| RRC Consent Form | Informed Consent | 01/12/2023 | 05/12/2023 |

\_\_\_\_\_\_


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

\_\_\_\_\_\_

\* \* \* Assent Background \* \* \*

#### 12. Assent Background

#### (Complete if applicable)

Assent Document: A form or script of the information that will be conveyed to the child about the study. In general, researcher must obtain the affirmative agreement of children ages seven years and older for their participation. Assent forms should be written at a level understandable to the child. If the study includes a broad age range of hildren, more than one assent form may be needed (i.e., an assent form suitable for a 17 year old is not usually suitable for a 7 year old child).

Assent Waiver: No child assent will be sought at all. This means that the IRB is asked to waive the requirement for child assent. Among other circumstances, this option is appropriate when the capability of the child to understand the research is too limited or when the research holds out a prospect of direct benefits that is important to the health or well-being of the child.

All minors must provide an affirmative consent to participate by signing a simplified assent form, unless the Investigator(s) provides evidence to the IRB that the minor subjects are not capable of assenting because of age, maturity, psychological state, or other factors.

Provide assent process background information, in the space below, for each Assent Form, Alteration Form (i.e., Cover Letter or Verbal Script), and Waiver.

\_\_\_\_\_\_


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

-----

#### \* \* \* HIPAA \* \* \*

#### 13. Health Insurance Portability and Accountability Act (HIPAA)

# If you are using PHI and this page is not active you must return to the General Checklist and check the box regarding the use of PHI in this research.

The HIPAA Privacy Rule establishes the right of an individual to authorize a covered entity, such as health plan, health care clearinghouse or health care provider, to use and disclose his/her Protected Health Information (PHI) for research purposes.

The Privacy Rule defines the elements of individual information that comprise PHI and establishes the conditions under which PHI may be used or disclosed by covered entities for research purposes. It also includes provisions to allow an individual's PHI to be disclosed or used in research without the person's authorization (i.e., IRB Waiver of HIPAA Requirement Authorization).

#### Is Your Research Covered by HIPAA's Privacy Rule? - Decision Tree

HIPAA Authorization Form

Waiver or Alteration of Authorization Form

Preparatory to Research Form

Limited Data Set/Data Use Agreement

Use and Disclosure of Decedents PHI without Authorization

Protected Health Information (PHI) is health information with one or more of the following identifiers. For more information see: http://privacyruleandresearch.nih.gov/clin\_research.asp or consult HIPAA Privacy Rule for Research

Research which involves the use of de-identified data is exempt from HIPAA requirements. In order to be de-identified data. NONE of the subject identifiers listed below can be collected, used, reviewed, recoded, accessed or disclosed.

Please review the following list and indicate if any of the information will be collected from any medical records for the purpose of this research project.

- 1 X Names
- 2. X Social Security Numbers
- 3. Telephone Numbers
- 4. All geographic subdivisions smaller than a state, including street address, city, county, precinct, zip code, and their equivalent geocodes, except for the initial three digits of a zip code, if according to the current publicly available data from the Bureau of the Census;
  - The geographic unit formed by combining all zip codes with the same three initial digits contains more than 20,000 people;
     and
  - ii. The initial three digits of a zip code for all such geographic units containing 20,000 or fewer people is changed to 000.
- 5. X All elements of dates (except year) for dates directly related to an individual, including birth date, admission date, discharge date, date of death; and all wages over 89 and all elements of dates (including year) indicative of such age, except that such ages and elements may be aggregated into a single category of age 90 or older.
- 6. Fax Numbers
- 7. Electronic Mail Addresses
- 8. Medical Record Numbers
  - You must attach a data collection sheet identifying the data points being collected from the MRN
- 9. Health Plan Beneficiary Numbers
- Account Numbers
- Certificate/License Numbers
- 12. Vehicle Identifiers and Serial Numbers, including License Plate Numbers
- 13. Device Identifiers and Serial Numbers
- 14. Web Universal Resource Locations (URLs)
- 15. Internet Protocol (IP) Address Numbers
- 16. Biometric Identifiers, including Finger and Voice Prints
- 17. Full Face Photographic Images and any Comparable Images


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

\_\_\_\_\_\_

18. Any other unique identifying number, character, or code (note this does not mean the unique code assigned by the Investigator(s) to code the research data)

\_\_\_\_\_\_

#### \* \* \* Potential Conflict of Interest \* \* \*

#### Potential Conflict of Interest

Conflict of Interest and the definitions related to the Conflict of Interest Policy and the following questions, please refer to the Help Screen.

#### Conflict of Interest: Please check Yes or No for each item below.

- a) Does the research involve a drug, device, or biological invented by you, an immediate family member or other Research Personnel?
- b) Is the research sponsored by an entity with which you, an immediate family member, or other Research Personnel have a paid consulting or advising relationship?
- **c)** Will you, members of your immediate family, or other Research Personnel receive special compensation or increased compensation if the research generates a favorable outcome?
- d) Will you, members of your immediate family, or other Research Personnel receive any money, gift or anything of monetary value above and beyond the actual costs of enrollment, conduct of the research, and reporting on the results, including, but not limited to, finders fees, referral fees, recruitment bonuses, and an enrollment bonus for reaching an accrual goal or similar types of payments?
- e) Do you, members of your immediate family or other Research Personnel have any other interests or relationships (including volunteer services) that might constitute a conflict of interest or an appearance of conflict of interest in connection with the research project?
- f) Will the payment you receive for services provided during the conduct of the research (e.g., investigator and Research Personnel time and tests) be inconsistent with fair market value for those services?

#### Significant Financial Interest: Please check Yes or No for each item below.

- g) Will you, your immediate family members or other Research Personnel receive salaries, royalties and/or other payments for services (e.g., consulting fees, honoraria, research design, management position, independent contractor, service on advisory or review committees, board membership seminars, lectures or teaching engagements when totaled together exceeded \$5,000 during the previous 12 months or are expected to exceed \$5,000 over the next 12 months)? This excludes reasonable costs of conducting the research, as specified in the research agreement.
- h) Do you, your immediate family members, or other Research Personnel hold any ownership interests including stocks, bonds, or stock options that exceed \$5,000 and/or that constitute more than a five percent (5%) ownership interest in the sponsoring organization? This does not include any interests held solely by reason of investment in a business by a mutual, pension or other institutional investment fund over which the investigator and/or his or her immediate family do not exercise day-to-day control of investment decisions.

If either g or h are Yes, is there a management plan in place?

If you have a management plan, is the COI being managed related to human subject research and/or this protocol?

#### Minimizing Risks and Disclosure to Subjects

- i) Have you disclosed any actual, potential or perceived conflicts of interest in the consent form? Research Personnel are required to disclose all such conflicts to all research participants in the research consent form.
- j) What steps, if any, have you taken or will you take to manage the conflict of interest and minimize the risks associated with any actual, potential or perceived conflicts of interest arising out of this research?

If you checked Yes to any statement (a-h, except f) above, please identify the research team member(s) below and provide details concerning the potential conflict of interest.

By submitting this form, you are attesting that you have read the The University of Notre Dame HRPP Policy on Conflict of Interest and agree to abide by its terms. You will update this disclosure form when new or changes in conflict of interest arise, and that you will comply with any conflict management plan required by the Institutional Review Board (IRB) to manage, reduce, or eliminate any actual or potential conflict of


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

\_\_\_\_\_

interest for the duration of the research.

\_\_\_\_\_

\* \* \* Attachments \* \* \*

#### 16. Attachments

Attach relevant documents here. These could include:

- Collaborating Investigator's IRB approval and approved documents
- Conflict of Interest information
- Debriefing Script; Grant/Sub-contract
- HIPAA Authorization Form from HIPAA-covered entity
- Interview/Focus Group Questions
- Investigator's Brochure
- Letters of Agreement/Cooperation from organizations who will help with recruitment
- Methodology section of associated Thesis or Dissertation project
- Questionnaires
- Radiation Control Office approval material
- Recruitment Material (e.g., flyers, email text, verbal scripts)
- Sponsor's Protocol; Surveys
- Other files associated with the protocol (you can upload most standard file formats: xls, pdf, jpg, tif, etc.)

Please be sure to attach all documents associated with your protocol. Failure to attach the files associated with the protocol may result in this protocol being returned to you for completion prior to being reviewed.

Students: Be sure to attach the Methods section of your thesis or dissertation proposal. If this protocol is associated with a grant proposal, please remember to attach your grant.

To update or revise any attachments, please delete the existing attachment and upload the revised document to replace it.

| Document Type | Document Name | Attached Date | Submitted Date |
|---|---|---|---|
| Other, supplemental information | CITI Basic & Research<br>Carla Exp 12.15.23 | 05/24/2021 | 05/24/2021 |
| Other, supplemental information | CITI Basic & Research<br>Chelsi Exp. 3.14.24 | 05/24/2021 | 05/24/2021 |
| Other, supplemental information | CITI Basic & Research<br>David Exp. 3.17.24 | 05/24/2021 | 05/24/2021 |
| Other, supplemental information | CITI Basic & Research<br>Juana Exp 6.8.22 | 05/24/2021 | 05/24/2021 |
| Other, supplemental information | CITI Basic & Research<br>Laurie Exp. 3.21.24 | 05/24/2021 | 05/24/2021 |
| Other, supplemental information | CITI Basic & Research<br>Mike Exp. 3.17.24 | 05/24/2021 | 05/24/2021 |
| Other, supplemental information | CITI Basic Casey Exp<br>9.18.22 | 05/24/2021 | 05/24/2021 |
| Other, supplemental information | CITI Research Casey Exp<br>9.17.24 | 05/24/2021 | 05/24/2021 |

e-Protocol


Protocol # 21-05-6633 Date Printed: 08/22/2023

Protocol Title: Recovery Resource Council - Veteran Incentives

Protocol Type: Protocol Submission Form

Date Submitted: 08/14/2023

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

-----

| Other, supplemental information | CITI Research Federico<br>04.12.21 | 05/24/2021 | 05/24/2021 |
|---|---|---|---|
| Other, supplemental information | Skira_CITICompletionCer tificate_April2021 | 05/24/2021 | 05/24/2021 |
| Explanatory diagram (Sequence of events) | RRC Enrollment Diagram 2020.09.15 | 05/24/2021 | 05/24/2021 |
| Questionnaires | RRC Intake Form for Consenting Clients | 05/24/2021 | 05/24/2021 |

\_\_\_\_\_

## \* \* \* Obligations \* \* \*

#### **Obligations**

#### The Principal Investigator of this study provides the following attestations:

- The eProtocol application submitted for this study is complete and accurate.
  - X The Principal Investigator has read and agrees to the above.
- The Principal Investigator has evaluated the protocol and determined that s/he has sufficient resources to conduct the study as submitted.
- The Principal Investigator will not begin the study until s/he has received notification of final determination of non-human subjects research.
  - X The Principal Investigator has read and agrees to the above.
- The Principal Investigator acknowledges his/her responsibility for the accuracy of all documents research personnel submit to the IRB on his/her behalf.
- The Principal Investigator will comply with all Research Compliance requests to report on the status of the study.
  - X The Principal Investigator has read and agrees to the above.

#### Non-Human Subjects research:

The Principal Investigator will not conduct research procedures outside of those described in the submission without prior review and approval.

#### · Exempt research:

The Principal Investigator will seek and obtain prior approval from the IRB for any modifications which may affect the Exempt status of the study.

#### Expedited/Full Board research:

The Principal Investigator will seek and obtain prior approval from the IRB for modifications to the study, including changes in procedures, consent forms, etc.

- X The Principal Investigator has read and agrees to the above.
- The Principal Investigator will promptly report any unexpected or otherwise significant adverse events or unanticipated problems or incidents that may occur in the course of this study.
- · The Principal Investigator will notify the IRB when his/her research has been completed or terminated.
  - X The Principal Investigator has read and agrees to abide by the above obligations.

The certification below should only be completed if this study has a student listed as Principal Investigator. Only the faculty member listed on the Personnel Information tab can check this box. No notification is sent to the Faculty Advisor, since the status of the protocol does not change until the form is submitted. Please contact the Faculty Advisor listed, and ask them to login to eProtocol using their own credentials. They will find this study on the first page, from which they should select "Edit" and review the submission. Once they approve, they can click on the box below, save the submission, and either submit or notify the student that the form can be submitted.

e-Protocol


Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

Protocol Submission Form **Protocol Type:** 

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

The Faculty Advisor has reviewed the protocol, finds the information to be complete and accurate, and agrees to serve as the responsible advisor for this protocol.

## \* \* \* Event History \* \* \*

#### **Event History**

| Date | Status | View Attachments | Letters |
|---|---|---|---|
| 05/14/2021 | NEW FORM CREATED | | |
| 05/24/2021 | NEW FORM<br>SUBMITTED | Y | |
| 06/09/2021 | NEW FORM PANEL<br>ASSIGNED | | |
| 06/10/2021 | NEW FORM PANEL<br>REASSIGNED | | |
| 06/10/2021 | NEW FORM<br>REVIEWER(S)<br>ASSIGNED | | |
| 08/05/2021 | NEW FORM SUBMITTED (CYCLE 1) - Application type switched to EXEMPT from EXPEDITED | Υ | |
| 08/16/2021 | NEW FORM<br>SUBMITTED (CYCLE 2) | Υ | |
| 09/09/2021 | NEW FORM<br>SUBMITTED (CYCLE 3) | Υ | |
| 09/09/2021 | NEW FORM APPROVED | Υ | Υ |
| 08/01/2022 | AMENDMENT 1 FORM<br>CREATED | | |
| 08/01/2022 | AMENDMENT 1 FORM<br>SUBMITTED | Υ | |
| 08/01/2022 | AMENDMENT 1 FORM<br>PANEL ASSIGNED | | |
| 08/01/2022 | AMENDMENT 1 FORM<br>REVIEWER(S)<br>ASSIGNED | | |
| 08/01/2022 | AMENDMENT 1 FORM SUBMITTED (CYCLE 1) | Υ | |
| 08/02/2022 | AMENDMENT 1 FORM<br>APPROVED | Υ | Υ |
| 01/12/2023 | AMENDMENT 2 FORM<br>CREATED | | |


Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

| 01/12/2023 | AMENDMENT 2 FORM SUBMITTED | Υ | |
|------------|---------------------------------------------|---|---|
| 01/12/2023 | AMENDMENT 2 FORM PANEL ASSIGNED | | |
| 01/12/2023 | AMENDMENT 2 FORM<br>REVIEWER(S)<br>ASSIGNED | | |
| 01/12/2023 | AMENDMENT 2 FORM SUBMITTED (CYCLE 1) | Υ | |
| 01/13/2023 | AMENDMENT 2 FORM<br>APPROVED | Υ | Υ |
| 05/12/2023 | AMENDMENT 3 FORM CREATED | | |
| 05/12/2023 | AMENDMENT 3 FORM SUBMITTED | Υ | |
| 05/15/2023 | AMENDMENT 3 FORM PANEL ASSIGNED | | |
| 05/15/2023 | AMENDMENT 3 FORM<br>REVIEWER(S)<br>ASSIGNED | | |
| 05/15/2023 | AMENDMENT 3 FORM APPROVED | Υ | Υ |
| 08/04/2023 | AMENDMENT 4 FORM CREATED | | |
| 08/04/2023 | AMENDMENT 4 FORM SUBMITTED | Υ | |
| 08/04/2023 | AMENDMENT 4 FORM PANEL ASSIGNED | | |
| 08/04/2023 | AMENDMENT 4 FORM<br>REVIEWER(S)<br>ASSIGNED | | |
| 08/04/2023 | AMENDMENT 4 FORM<br>APPROVED | Υ | Υ |
| 08/14/2023 | AMENDMENT 5 FORM CREATED | | |
| 08/14/2023 | AMENDMENT 5 FORM SUBMITTED | Υ | |
| 08/15/2023 | AMENDMENT 5 FORM PANEL ASSIGNED | | |
| 08/15/2023 | AMENDMENT 5 FORM<br>REVIEWER(S)<br>ASSIGNED | | |
| 08/15/2023 | AMENDMENT 5 FORM<br>APPROVED | Υ | Υ |


Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

Disclaimer: The generated PDF may not duplicate the original format completely. We do not warrant the accuracy of the changed format.

## \* \* \* Attached Document \* \* \*

| Document Name | Created Date |
|----------------------------------------------|--------------|
| CITI Basic & Research Carla Exp 12.15.23.pdf | 08/14/2023 |





Completion Date 15-Dec-2020 Expiration Date 15-Dec-2023 Record ID 39954756

This is to certify that:

## Carla Ervin

Has completed the following CITI Program course:

Not valid for renewal of certification through CME.

## **Human Research**

(Curriculum Group)

## Social & Behavioral Research

(Course Learner Group)

1 - Basic Course

(Stage)

Under requirements set by:

**University of Notre Dame** 



Verify at www.citiprogram.org/verify/?w89cd0e81-11c5-4936-9bca-b611b91c9bd9-39954756


Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

## \* \* \* Attached Document \* \* \*

| Document Name | Created Date |
|-----------------------------------------------|--------------|
| CITI Basic & Research Chelsi Exp. 3.14.24.pdf | 08/14/2023 |





Completion Date 15-Mar-2021 Expiration Date 14-Mar-2024 Record ID 40927479

This is to certify that:

## Chelsi Najera

Has completed the following CITI Program course:

**Human Research** 

(Curriculum Group)

Social & Behavioral Research

(Course Learner Group)

1 - Basic Course

(Stage)

Under requirements set by:

**University of Notre Dame** 

Not valid for renewal of certification through CME.



Verify at www.citiprogram.org/verify/?w9048c42a-ba89-4c5c-8b71-6726364bab80-40927479


Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

## \* \* \* Attached Document \* \* \*

| Document Name | Created Date |
|----------------------------------------------|--------------|
| CITI Basic & Research David Exp. 3.17.24.pdf | 08/14/2023 |





Completion Date 18-Mar-2021 Expiration Date 17-Mar-2024 Record ID 41282951

This is to certify that:

## David Ha

Has completed the following CITI Program course:

**Human Research** 

(Curriculum Group)

Social & Behavioral Research

(Course Learner Group)

1 - Basic Course

(Stage)

Under requirements set by:

**University of Notre Dame** 

Not valid for renewal of certification through CME.



Verify at www.citiprogram.org/verify/?w92f26b24-3bea-4c15-b557-098a05637885-41282951


Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

## \* \* \* Attached Document \* \* \*

| Document Name | Created Date |
|--------------------------------------------|--------------|
| CITI Basic & Research Juana Exp 6.8.22.pdf | 08/14/2023 |





Completion Date 09-Jun-2019 Expiration Date 08-Jun-2022 Record ID 31788674

This is to certify that:

Juana Garcia

Has completed the following CITI Program course:

Social & Behavioral Research - Basic/Refresher (Curriculum Group)

Social & Behavioral Research - Basic/Refresher (Course Learner Group)

1 - Basic Course

Under requirements set by:

**Texas Woman's University** 

(Stage)

**Collaborative Institutional Training Initiative** 

Verify at www.citiprogram.org/verify/?wa26b607c-0fc9-4853-aa37-31dc6006546f-31788674


Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

## \* \* \* Attached Document \* \* \*

| Document Name | Created Date |
|-----------------------------------------------|--------------|
| CITI Basic & Research Laurie Exp. 3.21.24.pdf | 08/14/2023 |




Completion Date 22-Mar-2021 Expiration Date 21-Mar-2024 Record ID 41682861

This is to certify that:

## **Laurie Mitchell**

Has completed the following CITI Program course:

**Human Research** 

(Curriculum Group)

Social & Behavioral Research

(Course Learner Group)

1 - Basic Course

(Stage)

Under requirements set by:

**University of Notre Dame** 

Not valid for renewal of certification through CME.



### **PROTOCOL Protocol Submission Form**

Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

| Document Name | Created Date |
|---------------------------------------------|--------------|
| CITI Basic & Research Mike Exp. 3.17.24.pdf | 08/14/2023 |





Completion Date 18-Mar-2021 Expiration Date 17-Mar-2024 Record ID 40926743

This is to certify that:

## Mike Fowler

Has completed the following CITI Program course:

Human Research

(Curriculum Group)

Social & Behavioral Research

(Course Learner Group)

1 - Basic Course

(Stage)

Under requirements set by:

**University of Notre Dame** 

Not valid for renewal of certification through CME.



Verify at www.citiprogram.org/verify/?w3b99398c-a561-42ce-9544-73c4b6d76497-40926743

### **PROTOCOL Protocol Submission Form**

Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

| Document Name | Created Date |
|----------------------------------|--------------|
| CITI Basic Casey Exp 9.18.22.pdf | 08/14/2023 |





Completion Date 19-Sep-2019 Expiration Date 18-Sep-2022 Record ID 33414625

This is to certify that:

## **Casey Gutierrez**

Has completed the following CITI Program course:

Social & Behavioral Research - Basic/Refresher

(Curriculum Group)

Social & Behavioral Research - Basic/Refresher

(Course Learner Group)

1 - Basic Course

(Stage)

Under requirements set by:

**Texas Woman's University** 

Not valid for renewal of certification through CME.



Verify at www.citiprogram.org/verify/?wffb99728-4fa3-4e5c-a797-4045d6a8e00b-33414625

### **PROTOCOL Protocol Submission Form**

Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

| Document Name | Created Date |
|-------------------------------------|--------------|
| CITI Research Casey Exp 9.17.24.pdf | 08/14/2023 |





Completion Date 19-Sep-2019 Expiration Date 17-Sep-2024 Record ID 27849103

This is to certify that:

## **Casey Gutierrez**

Has completed the following CITI Program course:

Social and Behavioral Responsible Conduct of Research

(Curriculum Group)

Social and Behavioral Responsible Conduct of Research

(Course Learner Group)

1 - RCR

(Stage)

Under requirements set by:

**Texas Woman's University** 

Not valid for renewal of certification through CME.



Verify at www.citiprogram.org/verify/?wc0bdffe4-ab18-4d5d-b4b9-3c9f3e869140-27849103

### **PROTOCOL Protocol Submission Form**

Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

| Document Name | Created Date |
|-------------------------------------|--------------|
| CITI Research Federico 04.12.21.pdf | 08/14/2023 |





Completion Date 12-Apr-2021 Expiration Date 11-Apr-2024 Record ID 41793667

This is to certify that:

## Federico Mendez

Has completed the following CITI Program course:

**Human Research** 

(Curriculum Group)

Social & Behavioral Research

(Course Learner Group)

1 - Basic Course

(Stage)

Under requirements set by:

**University of Notre Dame** 

Not valid for renewal of certification through CME.



Verify at www.citiprogram.org/verify/?wc9d49de3-ce8c-4cae-adfd-ab03037cf1b3-41793667

### **PROTOCOL Protocol Submission Form**

Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

| Document Name | Created Date |
|-----------------------------------------------|--------------|
| Skira_CITICompletionCertificate_April2021.pdf | 08/14/2023 |





Completion Date 09-Apr-2021 Expiration Date 08-Apr-2026 Record ID 28580198

This is to certify that:

# Meghan Skira

Has completed the following CITI Program course:

**Human Research** 

(Curriculum Group)

Social & Behavioral Research

(Course Learner Group)

2 - Refresher Course

(Stage)

Under requirements set by:

**University of Georgia** 

Not valid for renewal of certification through CME.



Verify at www.citiprogram.org/verify/?w25918bdb-db9a-4259-a1ee-b89cdbe5e6bc-28580198

### **PROTOCOL Protocol Submission Form**

Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

| Document Name | Created Date |
|---------------------------------------|--------------|
| RRC Enrollment Diagram 2020.09.15.pdf | 08/14/2023 |

### Recovery Resource Council (RRC) Study Enrollment



#### Notes:

- (1) Most clients are referred to the program through the Dallas-Fort Worth and Metroplex. Others are referred by veteran friendly agencies, word of mouth, and community partners.
- (2) Individuals who are eligible must be a veteran. They are assigned an intake session date and told to bring proof of their veteran ID to the intake session.
- (3) The veteran shows requested documentation, completes an intake form that collects demographic information, completes initial assessments, and a case is created for the individual. From here, veterans may give RRC their counseling recommendations (i.e. male/female counselor, etc). As a part of the standard intake process, the study will be introduced to the veteran and they will be asked if they would like to participate in the research study.

### **PROTOCOL Protocol Submission Form**

Protocol # 21-05-6633 Date Printed: 08/22/2023

**Protocol Title:** Recovery Resource Council - Veteran Incentives

**Protocol Type:** Protocol Submission Form

**Date Submitted:** 08/14/2023

**Important Note:** 

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

| Document Name | Created Date |
|---------------------------------------------|--------------|
| RRC Intake Form for Consenting Clients.docx | 08/14/2023 |



For official use only: \_\_\_\_\_\_

#### Providing hope, conquering addiction, healing families.

# **CLIENT INFORMATION**

| Name: | | Dat | e of Birth: _ | L | ast 4 SS#: | Gend | er: |
|---|---|---|---|---|---|---|---|
| \ddress: | | | | | | | |
| City: | | St | ate: | Zip: | Coun | ty: | |
| Email: | | | | | | | |
| | | , | | | <i>,</i> , , | | |
| 'hone: <u>( </u> | ) | ( | ) | | ( ) | | |
| hone: <u>(</u><br>Hon | | Cell | ) | | Work | | |
| Hon | ne | | | | Work | | |
| Hon<br>f you live in | ne | Cell<br>ty, <u>please circle c</u> | | | Work | | |
| Hon<br>f you live in | ne<br>n Tarrant Coun<br>thwest Tarran | Cell<br>ty, <u>please circle c</u> | one of the 3 | 7 areas with | Work<br>in the four reg | gions listed b | |
| Hon f you live in Nor Alliance | ne<br>n Tarrant Coun<br>thwest Tarran<br>Azle | Cell<br>ty, <u>please circle c</u><br>t County: | one of the 3 | <b>7 areas with</b><br>Carswell | Work in the four reg | gions listed b | <b>elow:</b><br>Haslet |
| Hon f you live in Nor Alliance ake Worth | ne<br>n Tarrant Coun<br>thwest Tarran<br>Azle | Cell<br>ty, <u>please circle o</u><br>t County:<br>Blue Moun<br>ver Oaks | one of the 3 | <b>7 areas with</b><br>Carswell | Work in the four reg | gions listed b | <b>elow:</b><br>Haslet |
| Hon f you live in Nor Alliance ake Worth | ne<br>n Tarrant Coun<br>thwest Tarran<br>Azle<br>Ri | Cell ty, please circle of t County: Blue Moun ver Oaks | one of the 3 | <b>7 areas with</b><br>Carswell<br>Sans | Mork in the four reg Fort Work som Park | gions listed b | <b>elow:</b><br>Haslet |
| Hon f you live in Nor Alliance ake Worth Nor Sedford | ne<br>n Tarrant Coun<br>thwest Tarran<br>Azle<br>Ri<br>theast Tarrant | Cell ty, please circle of t County: Blue Moun ver Oaks | one of the 37<br>d<br>Saginaw | <b>7 areas with</b><br>Carswell<br>Sans | Mork in the four reg Fort Work som Park | gions listed b<br>th<br>White | <b>elow:</b> Haslet Settlement |

| Arlington | Everman | Forest Hill | Fort Worth | Grand Prairie |
|---|---|---|---|---|
| Kennedale | Mansfield | | | |
| 4 | | | | |
| 4. Southwest Ta | rrant County: | | | |
| Benbrook | Crowley | Edgecliff | Fort Worth | Burleson |
| Were services easily a | ccessible? Yes | No | | |
| Are you or anyone in | your family in the milita | ry or a Veteran? Yes | No | |
| Affiliation to you (plea | ase circle): 1. Self. 2. Spo | ouse. 3. Child. 4. Parents | s. 5. Grandparents. 6. Si | gnificant other. |
| Current status (circle | <b>one):</b> Active. Discha | rged. Reserv | e. Retired. | |
| Primary race/ethnic g | roup in which you ident | ify yourself (please circle | e): | |
| 1. Caucasian/Anglo/Eu | ıropean 2. Black/Africa | n American 3. Hispani | c/Latin 4.Native Ame | rican 5. Asian 6 |
| East Indian 7. Alaska | an Native 8. Hawaiian N | Native/ Pacific Islander | 9. Mediterranean 10. | Middle Eastern |
| 11.Mixed Race/ethnic | ity | | | |
| What is your primary | language/dialect? | | | |
| Will you need translat | tion/interpretation servi | ces? | | |
| Do you have special co | ommunication needs? S | pecify: | | |
| Education (highest gra | ade completed): | | | |
| <b>Current employment:</b> | 1.Full-time2.Part-1 | time3.Temp4.Une | mployed5.Disabled _ | _6.Retired |
| What is your total hou | usehold size? Please incl | ude in this number any a | and all persons living in | your home full |
| time, as well as any po | erson who lives outside | the home but can be cla | imed as a dependent fo | r tax purposes. |
| (Example: a full-time | college student who reco | eive most or all their fina | ancial support from you | ): |
| Please check the option | on below where your an | nual household income | falls under: | |
| Less than 20,750 | _20,750-34,59934,60 | 0-55,34955,350+ | | |

| following: salary/wages, VA disabilit | | | ployment benefits, | retirement plan |
|---|---|---|---|---|
| child support, and alimony: | | <del></del> | | |
| Relationship Status (please check):6.Remarried7.Widowed | 1.Single | 2.Married | 4.Separated _ | 5.Divorced |
| Emergency Contact Information: | | | | |
| Name, number and relationship: | | | | |
| What is your goal for counseling? | | | | |
| Please indicate where I can leave a n | nessage (please | check): Hom | neCellWo | orkemail |
| Other specify: | | | | |
| How many months of Trade School o | or Business Coll | ege? | or Not Applica | ble: |
| If currently in school, what is your ac | cademic perforr | mance or GPA (gra | ade point average) | ? |
| So far, have you achieved your educ | ational goals? _ | 1. Yes or | 2. No | |
| If not in school, would you consider | attending schoo | ol in the future? _ | 1. Yes or | 2. No |
| If not in school, are you interested in | n an education r | eferral?1 | . Yes or2.N | lo |
| If yes, what are your needs? | | | | |
| Do you live with (please circle as ma | ny as apply): 1 | . Spouse/ Significa | ant Other 2 | 2.Children |
| 3.Parents | 4.Grandpare | ents | | |

| _ | _ | | |
|---|----|-----|-----|
| 5 | F٢ | iei | าds |

## 6. Multi-Family

| Spouse Name: | | | | |
|---|---|---|---|---|
| Dependent Names & Ages: | | | | |
| | | | | _ |
| Military Information | | | | |
| Military branch you are affiliated (please circle): | 1. Air Force | 2. Army | 3. Navy | 4. Marines |
| Other/ specify | | | | |
| Date Enlisted: | | | | |
| Date discharged: | Rank at dischar | ge: | | |
| Years you have served? | Unit of Deploy | ment: | | |
| List locations and year of all deployments: Locat | tion | | Ye | ar: |
| Location: | | Year: | | |
| Location: | | Year: | | |
| What was your job title/MOS? | | | | |

Circle experiences you may have had:

| 1. Active theater | 2. Hand-to-hand Combat | 3. Sexual abuse/Harassmo | ent 4. Non-Combat |
|---|---|---|---|
| Health Information | | | |
| Rate your health (plea | se checkmark):1.Excellent _ | 2.Good3.Average _ | 4.Fair5.Declining |
| Please circle if you are | : 1. Physically Disabled | 2.Mentally Disabled | 3. Physical + Mental Disability |
| List all current chronic | medical and/or mental illness o | diagnoses: | |
| Date of most recent p | rimary care physician exam? | | |
| Date of most recent sp | oecialist exam? | Type of Doctor? _ | |
| In the past 120-days h | ave you been admitted to an En | nergency Room; if so what | date? |
| What illness or condit | ion were you treated for in the | Emergency Room? | |
| In the past 120-days h | ave you been admitted to an in | patient hospital; if so what | date? |
| What illness or condit | ion(s) were you treated for inpa | tient? | |
| Are you experiencing | any pain now? YES NO | | |

If YES, please explain and rate your pain using the chart below:



| Please list all <i>prescribed</i> medications you are currently taking: |
|---|
| <u>Nutrition</u> |
| Do you have any allergies to food or medication? Specify: |
| Have you lost or gained more than 10 pounds in the last 6 months? YES NO |
| Have you experienced unintentional weight loss or gain? YES NO |
| Have you had a recent change in appetite? YES NO |
| Do you have any dental concerns (e.g., enamel erosion, cavities, tooth sensitivity/pain, etc.)? YES NO |
| Specify: |
| In terms of eating habits or behaviors, do you have any concerns (e.g., preoccupation with calories, induced vomiting, severe restriction of food intake, binge eating, etc.)? YES NO |
| Specify: |
| <u>Welfare</u> |
| Do you have any concerns about abuse, exploitation, or neglect of persons in the following categories: children, |
| people over the age of 65, or adults with disabilities? Please include yourself if applicable. YES NO Specify: |

| Has anyone limited your daily activities (e.g., food and water, medications, glasses or hearing aids, medical |
|---|
| care, etc.)? YES NO |
| Specify: |
| Has someone talked to you in a threatening way? YES NO |
| Specify: |
| Has someone forced you to give them money or sign strange papers? |
| YES NO |
| Specify: |
| Has anyone touched you without your consent or hit you? |
| YES NO |
| Specify: |
| Substance Use Information |
| Do you smoke?1.Yes or2.No If Yes, how many years have you chronically smoked? |
| If Yes, how many cigarettes do you smoke in a 24-hour period? |
| <u>Substances Use</u> |
| Please circle any and all illegal substances you have used in the past 12-months: |
| 1. Cocaine 2.Marijuana 3.Opioids 4.Stimulants 5.Hallucinogens |
| 6. Sedatives/Tranquilizers 7. Benzo(Xanax, Valium, etc) |

| How often do use these substances? | 1.Daily _ | 2.Weekly | 3.Monthly | 4.Rarely _ | 5.Never |
|---|---|---|---|---|---|
| 6. Mixed Use | | | | | |
| Age of 1 use? | | | | | |
| Do you have any legal problems arising | g from using | these substan | ces? | _1.Yes or | 2.No |
| Have you given up important social, we2.No | ork, or recre | ational activiti | es from substa | nce use? | 1.Yes or |
| Do you struggle with relapse?1. | Yes or | _2.No | | | |
| If yes, please explain: | | | | | |
| Do you have any family history of subs | tance abuse | ? If so please | explain: | | |
| <u>Alcohol</u> | | | | | |
| How often do you drink alcohol?1.D | Daily2.W | eekly3.№ | lonthly4. | Rarely5 | .Never |
| How many ounces of alcohol do you co | onsume each | n time you drin | ık? | | |
| Age of 1 use of alcohol? | | | | | |
| Have you given up important social, we | ork, or recre | ational activiti | ies from alcoho | l <b>use?</b> 1.Yes | or2.No |
| Do you have any legal problems arising | g from using | alcohol? | 1.Yes or | 2. | .No |
| Legal Issues | | | | | |
| Do you have any misdemeanors or felo | onies? If yes | please explain | : | | |

| Do you have any other current or past legal issues? If so please explain: |
|---|
| <u>Psychotherapy</u> |
| Considering how you are feeling today, as well as what you know about therapy/counseling generally, please answer the following three questions: |
| How upsetting do you expect the first two counseling/therapy sessions to be? |
| 1. Very upsetting2. Upsetting3. Neither upsetting, nor enjoyable4. Enjoyable5. Very Enjoyable |
| Compared to how you feel today, how do you think your symptoms will change after two counseling/therapsessions? |
| 1. Much worse2. Worse3. Slightly Worse4. No change5. Slightly better6. Better7. Much better |
| Compared to how you feel today, how do you think your symptoms will change after the full course of recommended counseling/therapy sessions? |
| 1. Much worse2. Worse3. Slightly Worse4. No change5. Slightly better6. Better7. Much better |

| Did someone recently suggest that you seek out counseling/therapy for help with your symptoms or is this |
|---|
| something you wanted to do yourself?1. Myself2. Someone else |
| If someone else suggested counseling/therapy, who was this person? |
| 1. Spouse/partner2. Other relative3. Employer4. Someone at the VA5. Other |
| How difficult will it be for you to attend counseling/therapy because of external factors like work, transportation, childcare, and so on? |
| 1. Very difficult2. Difficult3. Neither difficult, nor easy4. Easy5. Very easy |
| How often do your time and/or financial commitments change? |
| 1. Very often2. Often3. Occasionally4. Rarely5. Very rarely |
| Have you ever participated in any counseling/therapy programs?1.Yes or2.No |
| If Yes, please complete the following questions/statements about your last experience with counseling/therapy |
| The things I learned in counseling/therapy were |
| 1. Useless2. Somewhat beneficial3. Beneficial4. Very Beneficial |
| I found my time with the counselor/therapist to be |
| 1. Very upsetting2. Upsetting3. Neither upsetting, nor enjoyable4. Enjoyable5. Very Enjoyable |
| Over the course of treatment, my symptoms became |
| 1. Much worse2. Worse3. No change4. Better5. Much better |

| What was it, if anything, that did not work? |
|---|
| Did you attend all the recommended sessions offered/suggested/ or prescribed?1.Yes or2. No |
| How many sessions did you attend before stopping? |
| Are you <u>currently</u> receiving mental health counseling/therapy from any other sources?1. Yes or2. No |
| What are your preferences for counseling? |
| 1. Individual 2.Couples 3.Family 4.Play Therapy 5.Groups |
| Does religion or spirituality play a role in your life?1.Yes or2. No |
| If yes, in what way? |
| <u>Preferences</u> |
| The following questions regard your preferences over various financial payments. None of the questions have a "correct" answer; your answer should be based on your opinion. These questions are also purely hypothetical. You will not win or lose any real money by answering. |
| Suppose you have won a prize of \$500, which you can claim immediately. However, if you choose to wait, you will receive a prize that is larger than \$500. Please complete the following: |
| If you offer me at least \$ in <u>one week</u> , I'll wait to claim this larger amount; offer me less and I'll take the \$500 now. |

| If you offer me at l | east \$ in <u>si</u> | x weeks, I'll wait to claim this larger amount; offer me less and I'll take the |
|---|---|---|
| \$500 now. | | |
| | | ng game, where you are paid one amount of money if the coin lands on s on tails. Prior to the game, you are allowed to <u>choose one</u> from the |
| following sets of p | rizes, where the d | ollar amount in the "heads" column is your winnings if the coin lands on |
| heads and the doll | ar amount in the | "tails" column is your winnings if the coin lands on tails. |
| Please mark the <u>or</u> | Please mark the <u>one set of prizes</u> you would choose: | |
| Heads | Tails | |
| \$500 | \$500 | |
| \$430 | \$640 | |
| \$360 | \$785 | |
| \$285 | \$930 | |
| \$215 | \$1070 | |
| \$35 | \$1250 | |
| Section for Child or | Youth Clients On | ly |
| If this form is for a | child or youth clie | ent (under the age of 18), please complete the following: |
| What is the legal cu | ıstody status? | |
| Please identify any | legal guardian(s) <sub>-</sub> | |
| In the past month, | how much of a pro | oblem has your child had with nutrition? |
| 1. Almost Alway | /s2. Often | 3. Sometimes4. Almost Never5.Never |

| "I hereby certify that the above statements are true and a false statement may disqualify me for grant-funded s | nd correct to the best of my knowledge. I understand that services." |
|---|---|
| Client and/or Parent/Guardian Signature | Date |